CLINICAL TRIAL: NCT03912194
Title: Early Withdrawal Exposure and Negative Affect Withdrawal (NAW) Regulation Training for Smoking Cessation
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Peter Hendricks, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 000522656
Record Dates: First submitted 2019-04-05; First posted 2019-04-11 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Tobacco Dependence
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Early Withdrawal Exposure plus NAW Regulation Training (Experimental): The development, application, modification, and repeated practice of individualized withdrawal regulation strategies (e.g., behavioral and cognitive strategies for allaying withdrawal symptoms) across the first 4 hours of abstinence over 4 separate sessions.
  Interventions: Behavioral: cognitive-behavioral withdrawal regulation strategies; Behavioral: early withdrawal exposure
- Early Withdrawal Exposure plus Relaxation Control Training (Active Comparator): The development, application, modification, and repeated practice of relaxation strategies across the first 4 hours of abstinence over 4 separate sessions.
  Interventions: Behavioral: relaxation strategies; Behavioral: early withdrawal exposure
- NAW Regulation Training Only (Active Comparator): The development, application, modification, and repeated practice of individualized withdrawal regulation strategies (e.g., behavioral and cognitive strategies for allaying withdrawal symptoms) over 4 separate sessions involving smoking as usual.
  Interventions: Behavioral: cognitive-behavioral withdrawal regulation strategies
- Relaxation Control Training Only (Active Comparator): The development, application, modification, and repeated practice of relaxation strategies over 4 separate sessions involving smoking as usual.
  Interventions: Behavioral: relaxation strategies

INTERVENTIONS:
Behavioral: cognitive-behavioral withdrawal regulation strategies — Participants will generate and refine individualized withdrawal regulation strategies with the aid of a therapist
  Arms: Early Withdrawal Exposure plus NAW Regulation Training; NAW Regulation Training Only
Behavioral: relaxation strategies — Participants will generate and refine relaxation techniques with the aid of a therapist
  Arms: Early Withdrawal Exposure plus Relaxation Control Training; Relaxation Control Training Only
Behavioral: early withdrawal exposure — Exposure to the first 4 hours of abstinence across 4 separate sessions
  Arms: Early Withdrawal Exposure plus NAW Regulation Training; Early Withdrawal Exposure plus Relaxation Control Training

SUMMARY:
Smoking remains the single most preventable cause of morbidity and mortality in the United States, accounting for approximately half a million deaths every year. The current study will investigate the efficacy and mechanisms of change of a novel smoking cessation intervention. The current study will thus provide essential information regarding a treatment that has the potential to enhance the efficacy of existing smoking cessation interventions, thereby having a beneficial impact on the public health of the United States.

DETAILED DESCRIPTION:
Cigarette smoking remains the single most preventable cause of mortality and morbidity in the United States. Long-term abstinence rates for even the most rigorous of smoking cessation treatments range between 20% and 35%. It is therefore essential that research continue to investigate novel smoking cessation interventions. Leading contemporary theories of addiction motivation posit that the escape or avoidance of negative affect withdrawal (NAW) symptoms (e.g., anger, anxiety, and depression/sadness) constitutes a strong motivational basis for cigarette smoking and plays a critical role in relapse to cigarette use. However, whereas NAW symptoms appear to exert a powerful influence on smoking cessation treatment outcome, smoking cessation interventions may exert only modest effects on NAW symptoms. Accordingly, it has been proposed that smoking cessation interventions may be augmented by aiding smokers in the practice of NAW regulation strategies. The primary goal of this investigation is to evaluate an early withdrawal exposure plus NAW regulation training intervention for smoking cessation. Specific aims include evaluating the efficacy of the treatment components and investigating potential mediators and moderators of the treatment components. Participants will be adult smokers (N = 400) of at least 5 cigarettes per day with the intention to quit smoking. Using a factorial design, participants will be randomized to early withdrawal exposure (yes vs. no) and behavioral intervention (NAW regulation training vs. relaxation control training), resulting in four distinct conditions. The investigator's primary hypothesis is that early withdrawal exposure plus NAW regulation training will produce higher rates of seven-day point-prevalence abstinence at 1, 3, and 6 months after end-of-treatment, suggesting a synergistic (i.e., non-additive) effect of the two intervention components. Mediators (e.g., in-session withdrawal symptoms) and moderators (e.g., demographic characteristics, tobacco dependence) will be investigated via established analyses. These data will advance the experimental intervention with a focus on targeting mechanisms of change as well as participant characteristics to which the intervention may be tailored. The experimental intervention described in the current proposal has the potential to ultimately enhance the efficacy of existing smoking cessation interventions and will therefore contribute uniquely to the field.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* smoke at least 5 cigarettes per day
* Expired breath carbon monoxide (CO) reading of at least five parts per million
* report the intention to quit
* reside in the Birmingham area with no plan to relocate outside of the area in the next 6 months
* access to a telephone

Exclusion Criteria:

* inability to speak English
* presence of a condition that contraindicates use of the nicotine patch
* presence of conditions that might interfere with compliance with the protocol or greatly complicate treatment
* any acutely life-threatening disease
* concurrent participation in a formal treatment program for smoking cessation
* current use of any pharmacotherapy for smoking cessation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-24 (Estimated)

PRIMARY OUTCOMES:
Smoking cessation as evaluated by self-reported, biochemically-confirmed seven-day point-prevalence abstinence | 1 month after end-of-treatment
  Self reported abstinence from smoking ("no smoking, not even a puff) in the past seven days, biochemically confirmed by a breath carbon monoxide reading of 3 or less
Smoking cessation as evaluated by self-reported, biochemically-confirmed seven-day point-prevalence abstinence | 3 months after end-of-treatment
  Self reported abstinence from smoking ("no smoking, not even a puff) in the past seven days, biochemically confirmed by a breath carbon monoxide reading of 3 or less
Smoking cessation as evaluated by self-reported, biochemically-confirmed seven-day point-prevalence abstinence | 6 months after end-of-treatment
  Self reported abstinence from smoking ("no smoking, not even a puff) in the past seven days, biochemically confirmed by a breath carbon monoxide reading of 3 or less

SECONDARY OUTCOMES:
Cessation milestones as determined by the Timeline Followback Interview | 1 month after end-of-treatment
  1) Was initial abstinence achieved (was there any day of non-smoking within the first two weeks after the quit date; yes or no)?; 2) latency to lapse (number of days to the first cigarette after the quit day); 3) was there a progression from lapse to relapse (defined as seven consecutive days of smoking; yes or no)?
Cessation milestones as determined by the Timeline Followback Interview | 3 months after end-of-treatment
  1) latency to lapse (number of days to the first cigarette after the quit day); 2) was there a progression from lapse to relapse (defined as seven consecutive days of smoking; yes or no)?
Cessation milestones as determined by the Timeline Followback Interview | 6 months after end-of-treatment
  1) latency to lapse (number of days to the first cigarette after the quit day); 2) was there a progression from lapse to relapse (defined as seven consecutive days of smoking; yes or no)?
Physical tobacco dependence | 1 month after end-of-treatment
  Tobacco dependence as measured by the Fagerstrom Test of Cigarette Dependence (FTCD). The FTCD is a widely used 9-item measure of physical dependence. FTCD scores, computed from the sum of the items, range from 0 to 10, with greater scores indicating greater dependence.
Physical tobacco dependence | 3 months after end-of-treatment
  Tobacco dependence as measured by the Fagerstrom Test of Cigarette Dependence (FTCD). The FTCD is a widely used 9-item measure of physical dependence. FTCD scores, computed from the sum of the items, range from 0 to 10, with greater scores indicating greater dependence.
Physical tobacco dependence | 6 months after end-of-treatment
  Tobacco dependence as measured by the Fagerstrom Test of Cigarette Dependence (FTCD). The FTCD is a widely used 9-item measure of physical dependence. FTCD scores, computed from the sum of the items, range from 0 to 10, with greater scores indicating greater dependence.
Motivational tobacco dependence | 1 month after end-of-treatment
  Tobacco dependence as measured by the and the Wisconsin Inventory of Smoking Dependence Motives (WISDM) questionnaire. The WISDM-68 is a 68-item measure designed to assess dependence as a motivational state on 13 subscales: Affiliative Attachment, Automaticity, Loss of Control, Behavioral Choice, Cognitive Enhancement, Craving, Cue Exposure, Negative Reinforcement, Positive Reinforcement, Social and Environmental Goads, Taste and Sensory Properties, Tolerance, and Weight Control. Scores on each subscale, computed from the mean of their respective items, range from 1 to 7, with greater scores indicating greater dependence.
Motivational tobacco dependence | 3 months after end-of-treatment
  Tobacco dependence as measured by the and the Wisconsin Inventory of Smoking Dependence Motives (WISDM) questionnaire. The WISDM-68 is a 68-item measure designed to assess dependence as a motivational state on 13 subscales: Affiliative Attachment, Automaticity, Loss of Control, Behavioral Choice, Cognitive Enhancement, Craving, Cue Exposure, Negative Reinforcement, Positive Reinforcement, Social and Environmental Goads, Taste and Sensory Properties, Tolerance, and Weight Control. Scores on each subscale, computed from the mean of their respective items, range from 1 to 7, with greater scores indicating greater dependence.
Motivational tobacco dependence | 6 months after end-of-treatment
  Tobacco dependence as measured by the and the Wisconsin Inventory of Smoking Dependence Motives (WISDM) questionnaire. The WISDM-68 is a 68-item measure designed to assess dependence as a motivational state on 13 subscales: Affiliative Attachment, Automaticity, Loss of Control, Behavioral Choice, Cognitive Enhancement, Craving, Cue Exposure, Negative Reinforcement, Positive Reinforcement, Social and Environmental Goads, Taste and Sensory Properties, Tolerance, and Weight Control. Scores on each subscale, computed from the mean of their respective items, range from 1 to 7, with greater scores indicating greater dependence.
Withdrawal symptoms | 1 month after end-of-treatment
  Withdrawal symptoms as measured by the 28-item Wisconsin Smoking Withdrawal Scale (WSWS). The WSWS measures smoking withdrawal symptoms on 7 subscales: Anger, Anxiety, Concentration, Craving, Hunger, Sadness, and Sleep Difficulty. Scores on each subscale, computed from the mean of their respective items, range from 0 to 4, with greater scores indicating greater withdrawal.
Withdrawal symptoms | 3 months after end-of-treatment
  Withdrawal symptoms as measured by the 28-item Wisconsin Smoking Withdrawal Scale (WSWS). The WSWS measures smoking withdrawal symptoms on 7 subscales: Anger, Anxiety, Concentration, Craving, Hunger, Sadness, and Sleep Difficulty. Scores on each subscale, computed from the mean of their respective items, range from 0 to 4, with greater scores indicating greater withdrawal.
Withdrawal symptoms | 6 months after end-of-treatment
  Withdrawal symptoms as measured by the 28-item Wisconsin Smoking Withdrawal Scale (WSWS). The WSWS measures smoking withdrawal symptoms on 7 subscales: Anger, Anxiety, Concentration, Craving, Hunger, Sadness, and Sleep Difficulty. Scores on each subscale, computed from the mean of their respective items, range from 0 to 4, with greater scores indicating greater withdrawal.
Abstinence-related expectancies | 1 month after end-of-treatment
  Abstinence-related expectancies as measured by the 55-items Smoking Abstinence Questionnaire (SAQ). The SAQ measures expectancies for abstinence from smoking on 10 subscales: Withdrawal, Social Improvement/Non-smoker Identity, Adverse Outcomes, Treatment Effectiveness, Common Reasons, Barriers to Treatment, Social Support, Optimistic Outcomes, Coffee Use, and Weight Gain. Scores on each subscale, computed from the mean of their respective items, range from 0 to 6, with greater scores reflecting stronger expectancies.
Abstinence-related expectancies | 3 months after end-of-treatment
  Abstinence-related expectancies as measured by the 55-item Smoking Abstinence Questionnaire (SAQ). The SAQ measures expectancies for abstinence from smoking on 10 subscales: Withdrawal, Social Improvement/Non-smoker Identity, Adverse Outcomes, Treatment Effectiveness, Common Reasons, Barriers to Treatment, Social Support, Optimistic Outcomes, Coffee Use, and Weight Gain. Scores on each subscale, computed from the mean of their respective items, range from 0 to 6, with greater scores reflecting stronger expectancies.
Abstinence-related expectancies | 6 months after end-of-treatment
  Abstinence-related expectancies as measured by the 55-item Smoking Abstinence Questionnaire (SAQ). The SAQ measures expectancies for abstinence from smoking on 10 subscales: Withdrawal, Social Improvement/Non-smoker Identity, Adverse Outcomes, Treatment Effectiveness, Common Reasons, Barriers to Treatment, Social Support, Optimistic Outcomes, Coffee Use, and Weight Gain. Scores on each subscale, computed from the mean of their respective items, range from 0 to 6, with greater scores reflecting stronger expectancies.
Thoughts about abstinence | 1 month after end-of-treatment
  Motivation to quit, expected difficulty quitting, and confidence in one's ability to quit are measured by one item each by the Thoughts About Abstinence (TAA) questionnaire. Scores on each item range from 1 to 10, with greater scores indicating greater motivation to quit, expected difficulty quitting, and confidence in one's ability to quit, respectively.
Thoughts about abstinence | 3 months after end-of-treatment
  Motivation to quit, expected difficulty quitting, and confidence in one's ability to quit are measured by one item each by the Thoughts About Abstinence (TAA) questionnaire. Scores on each item range from 1 to 10, with greater scores indicating greater motivation to quit, expected difficulty quitting, and confidence in one's ability to quit, respectively.
Thoughts about abstinence | 6 months after end-of-treatment
  Motivation to quit, expected difficulty quitting, and confidence in one's ability to quit are measured by one item each by the Thoughts About Abstinence (TAA) questionnaire. Scores on each item range from 1 to 10, with greater scores indicating greater motivation to quit, expected difficulty quitting, and confidence in one's ability to quit, respectively.
Intolerance for smoking abstinence discomfort | 1 month after end-of-treatment
  Intolerance for smoking abstinence discomfort, as measured by the 17-tem Intolerance for Smoking Abstinence Discomfort Questionnaire (IDQ-S). The IDQ-S assesses the inability to tolerate smoking abstinence discomfort on two subscales: Withdrawal Intolerance and Lack of Cognitive Coping. Scores on each subscale, computed from the mean of their respective items, range from 1 to 5, with greater scores indicating greater inability to tolerate abstinence.
Intolerance for smoking abstinence discomfort | 3 months after end-of-treatment
  Intolerance for smoking abstinence discomfort, as measured by the 17-item Intolerance for Smoking Abstinence Discomfort Questionnaire (IDQ-S). The IDQ-S assesses the inability to tolerate smoking abstinence discomfort on two subscales: Withdrawal Intolerance and Lack of Cognitive Coping. Scores on each subscale, computed from the mean of their respective items, range from 1 to 5, with greater scores indicating greater inability to tolerate abstinence.
Intolerance for smoking abstinence discomfort | 6 months after end-of-treatment
  Intolerance for smoking abstinence discomfort, as measured by the 17-item Intolerance for Smoking Abstinence Discomfort Questionnaire (IDQ-S). The IDQ-S assesses the inability to tolerate smoking abstinence discomfort on two subscales: Withdrawal Intolerance and Lack of Cognitive Coping. Scores on each subscale, computed from the mean of their respective items, range from 1 to 5, with greater scores indicating greater inability to tolerate abstinence.

CONTACTS AND LOCATIONS:
Locations (1):
- Ryals Public Health Building, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No